CLINICAL TRIAL: NCT05437965
Title: National Multicenter Cohort Registry Study of Rapid rEcurrences of Coronary Unexplained In-stent Restenosis
Acronym: RECUR Registry
Status: Recruiting | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Chinese Academy of Medical Sciences, Fuwai Hospital (Other); The First Hospital of Jilin University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Kefei Dou, MD, Director of the Department of Internal Medicine, China National Center for Cardiovascular Diseases
Other Study IDs: 2021-ZX50
Record Dates: First submitted 2022-06-24; First posted 2022-06-29 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Coronary Artery Disease; Arteritis; In-Stent Stenosis (Restenosis) of Coronary Artery Stent
Keywords: coronary arteritis; biomarker; inflammation
MeSH Terms: conditions — Coronary Artery Disease; Arteritis; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Rapid rEcurrences of Coronary Unexplained in-stent Restenosis (RECUR)
  Interventions: Other: Treatment made by experienced clinicians

INTERVENTIONS:
Other: Treatment made by experienced clinicians — Treatment made by experienced clinicians

SUMMARY:
This project aims to establish a clinical cohort and diagnostic assessment framework by conducting a national multicenter cohort registry study. Through the collection of patients' clinical characteristics, it will achieve the registration, management, follow-up, and analysis of patients with Rapid rEcurrences of Coronary Unexplained in-stent Restenosis (RECUR).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Patients meeting the diagnostic criteria for Rapid rEcurrences of Coronary Unexplained in-stent Restenosis (RECUR);
3. Patients fully informed about the trial procedures who provide written informed consent.

Exclusion Criteria:

1. Patients presenting with any of the following:

   * Other severe comorbidities (e.g., malignant tumors, heart failure) with a life expectancy <12 months;

     * Known autoimmune/rheumatic diseases including systemic lupus erythematosus, Takayasu arteritis, Behçet's disease, polyarteritis nodosa, Wegener granulomatosis (granulomatosis with polyangiitis), eosinophilic arteritis, giant cell arteritis, rheumatoid arthritis, or IgG4-related disease;

       * Variant angina (Prinzmetal's angina);

         * Coronary artery dissection;

           * Thrombophilia;

             * Stent underexpansion.
2. Presence of psychiatric disorders;
3. Known inability to complete expected study follow-up for any reason;
4. Patients deemed ineligible for enrollment by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who meet the definition of Rapid rEcurrences of Coronary Unexplained in-stent Restenosis (RECUR), that is, patients who have undergone myocardial infarction or target vessel-related revascularization ≥3 times due to coronary artery stenosis in the past year after coronary stent implantation and standard coronary heart disease conventional treatment (complete revascularization and optimal medical therapy), excluding common risk factors for coronary artery restenosis and known rheumatic autoimmune diseases, systemic vasculitis, etc.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-06-03 (Actual); Primary Completion 2035-04-01 (Estimated); Study Completion 2035-04-01 (Estimated)

PRIMARY OUTCOMES:
Target vessel failure | 10 year
  Time to the incidence of target vessel failure, a composite of cardiovascular death, target vessel-related myocardial infarction, and target vessel-related revascularization.

CONTACTS AND LOCATIONS:
Locations (1):
- Jia Lei, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Study protocol, clinical study report can be shared.